CLINICAL TRIAL: NCT02011113
Title: A Phase 2, Multicenter, Single-arm, Open-label Study in Japan to Evaluate the Efficacy and Safety of Pomalidomide (CC-4047) in Combination With Dexamethasone in Subjects With Relapsed and Refractory Multiple Myeloma
Brief Title: Japanese Phase 2 Study to Evaluate the Efficacy and Safety of Pomalidomide in Subjects With Relapsed and Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-4047-MM-011
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Results first posted 2015-11-10 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-09

CONDITIONS: Multiple Myeloma
Keywords: Pomalidomide,; CC-4047,; Dexamethasone,; Relapsed and refractory multiple myeloma,; phase 2
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pomalidomide plus dexamethasone (Experimental)
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Pomalidomide — 4 mg oral pomalidomide once daily Days 1-21 of each 28-day cycle
  Other Names: CC-4047
Drug: Dexamethasone — 40 mg or 20 mg oral dexamethasone once daily on Days 1, 8, 15, 22 of each 28-day cycle
  Other Names: LenaDex

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of pomalidomide in combination with dexamethasone in subjects with relapsed and refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* 1. Must be ≥ 20 years of age at the time of signing the informed consent document.

  2. The subject must understand and voluntarily sign an informed consent document before any study related assessments/procedures are conducted.

  3. Must be able to adhere to the study visit schedule and other protocol requirements.

  4. Have a documented diagnosis of multiple myeloma and have relapsed and refractory disease. Subjects must have received at least 2 prior therapies. Subjects must have relapsed after having achieved at least stable disease for at least one cycle of treatment to at least one prior regimen and then developed progressive disease(PD). Subjects must also have documented evidence of progressive disease(PD) during or within 60 days (measured from the end of the last cycle) of completing treatment with the last antimyeloma drug regimen used just prior to study entry (refractory disease).

  5. Subjects must have undergone prior treatment with at least 2 cycles of lenalidomide and at least 2 cycles of bortezomib (either in separate regimens or within the same regimen).

  6. Subjects must have documented diagnosis of multiple myeloma and have measurable disease (serum M-protein ≥ 0.5 g/dL or urine M-protein ≥ 200 mg/24 hours).

  7. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2.

  8.Must agree to comply to pomalidomide Pregnancy Prevention Risk Management Plan.

Exclusion Criteria:

* 1. Pregnant or breastfeeding females 2. Hypersensitivity to thalidomide, lenalidomide, or dexamethasone 3. ≥ Grade 3 rash during prior thalidomide or lenalidomide therapy 4. Subjects unable or unwilling to undergo antithrombotic prophylactic treatment will not be eligible to participate in this study 5. Any of the following laboratory abnormalities:

  * Absolute neutrophil count < 1,000/µL
  * Platelet count < 75,000/µL for subjects in whom < 50% of bone marrow nucleated cells are plasma cells; or a platelet count < 30,000/µL for subjects in whom ≥ 50% of bone marrow nucleated cells are plasma cells
  * Creatinine Clearance < 45 mL/min according to Cockcroft-Gault formula

Cockcroft-Gault estimation of Creatinine Clearance:

* Corrected serum calcium > 14 mg/dL (> 3.5 mmol/L)
* Hemoglobin < 8 g/dL (< 4.9 mmol/L; prior Red blood cell transfusion or recombinant human erythropoietin use is permitted)
* Serum glutamic oxaloacetic transaminase(SGOT)/aspartate aminitransferase(AST) or serum glutamic pyruvic transaminase(SGPT)/alanine aminotransferase(ALT) > 3.0 x upper limit of normal(ULN)
* Serum total bilirubin > 2.0 mg/dL (34.2 μmol/L); or ≥ 3.0 x upper limit of normal (ULN) for subjects with hereditary benign hyperbilirubinemia.

  6. Subjects with any one of the following:
* Congestive heart failure (New York Heart Association Class III or IV)
* Myocardial infarction within 12 months prior to starting study treatment
* Unstable or poorly controlled angina pectoris, including Prinzmetal variant angina pectoris 7. Peripheral neuropathy ≥ Grade 2. 8. Prior history of malignancies, other than multiple myeloma, unless the subject has been free of the disease for ≥ 5 years. Exceptions include the following:
* Basal or Squamous cell carcinoma of the skin
* Carcinoma in situ of the cervix or breast
* Incidental histologic finding of prostate cancer (TNM stage of T1a or T1b) 9. Known infection with human immunodeficiency virus (HIV) antibody positive, hepatitis B virus surface antigen (HBsAg) positive or hepatitis C virus antibody (HCVAb) positive. If negative for hepatitis B virus surface antigen (HBsAg) but hepatitis B core antibody (HBcAb) and/or hepatitis B surface antibody (HBsAb) positive status, a hepatitis B virus DNA test will be performed and if positive the subject will be excluded.

  10. Incidence of gastrointestinal disease that may significantly alter the absorption of pomalidomide.

  11. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.

  12. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.

  13. Any condition that confounds the ability to interpret data from the study. 14. Previous therapy with pomalidomide. 15. Use of any investigational agents within 28 days or 5 half-lives (whichever is longer) of treatment.

  16. Subjects with conditions requiring chronic steroid or immunosuppressive treatment, such as rheumatoid arthritis, multiple sclerosis, and lupus, which likely need additional steroid or immunosuppressive treatments in addition to the study treatment. Includes subjects receiving corticosteroids (> 10 mg/day of prednisone or equivalent) within 3 weeks prior to enrollment.

  17. Subjects who received any of the following within the last 14 days of initiation of study treatment:
* Plasmapheresis
* Major surgery (kyphoplasty is not considered major surgery)
* Radiation therapy
* Use of any antimyeloma drug therapy. 18. Subjects who received an allogeneic bone marrow or allogeneic peripheral blood stem cell transplant less than 12 months prior to initiation of study treatment and who have not discontinued immunosuppressive treatment for at least 4 weeks prior to initiation of study treatment and are currently dependent on such treatment.

  19. Subjects who are planning for or who are eligible for stem cell transplant.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-12; Primary Completion 2014-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toru Sasaki, Director, Study Director — Celgene K.K.
Locations (11):
- Japan (11):
  - Celgene Trial Site, Nagoya, Aichi-ken
  - Celgene Trial Site, Kamogawa, Chiba
  - Celgene Trial Site, Fukuoka, Fukuoka
  - Celgene Trial Site, Hiroshima, Hiroshima
  - Celgene Trial Site, Mito, Ibaragi
  - Celgene Trial Site, Isehara, Kanagawa
  - Celgene Trial Site, Kyoto, Kyoto
  - Celgene Trial Site, Niigata, Niigata
  - Celgene Trial Site, Okayama, Okayama-ken
  - Celgene Trial Site, Osaka, Osaka
  - Celgene Trial Site, Tokyo, Tokyo

REFERENCES:
- [Derived] Ichinohe T, Kuroda Y, Okamoto S, Matsue K, Iida S, Sunami K, Komeno T, Suzuki K, Ando K, Taniwaki M, Tobinai K, Chou T, Kaneko H, Iwasaki H, Uemura C, Tamakoshi H, Zaki MH, Doerr T, Hagiwara S. A multicenter phase 2 study of pomalidomide plus dexamethasone in patients with relapsed and refractory multiple myeloma: the Japanese MM-011 trial. Exp Hematol Oncol. 2016 Apr 18;5:11. doi: 10.1186/s40164-016-0040-7. eCollection 2015. PMID 27096106

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All study participants who were on pomalidomide were transferred to the post-marketing study and continued the study treatment when pomalidomide became commercially available.
Pre-assignment Details: Treatment phase discontinuation occurred when a participant had confirmed progressive disease, development of unacceptable toxicity, voluntary withdrawal or met other criteria for treatment discontinuation.
Groups:
- Pomalidomide Plus Dexamethasone: Pomalidomide 4 mg by mouth (PO) daily (QD) on Days 1-21 of each 28-day cycle. Dexamethasone 40 mg PO once daily on Days 1, 8, 15, 22 of each 28-day cycle for those who are ≤ 75 years of age Dexamethasone 20 mg PO once daily on Days 1, 8, 15, 22 of each 28-day cycle for those who are > 75 years of age
Period: Overall Study
Arm/Group | Pomalidomide Plus Dexamethasone
Started | 36
Completed | 0 (Completed = participants with progressive disease were considered as completed.)
Not Completed | 36
Not completed — Adverse Event | 4
Not completed — Disease Progression (DP) | 16
Not completed — Death | 1
Not completed — Insufficient effect of Pomalidomide | 1
Not completed — Investigator's judgement- DP | 3
Not completed — Study terminated by sponsor | 11

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received at least one dose of study medication
Groups:
- Pomalidomide Plus Dexamethasone: Pomalidomide: 4 mg oral pomalidomide once daily Days 1-21 of each 28-day cycle Dexamethasone: 40 mg or 20 mg oral dexamethasone once daily on Days 1, 8, 15, 22 of each 28-day cycle
Arm/Group | Pomalidomide Plus Dexamethasone
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: years] | 64.5 [43 to 78]
Age, Customized [Number; unit: participants]
  ≤ 75 Years Old | 32
  > 75 Years Old | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 36
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Time from first diagnosis [Median (Full Range); unit: years] | 4.65 [0.6 to 21.1]
Durie-Salmon Multiple myeloma staging at screening [Number; unit: participants] — Stages are: Stage I: Hemoglobin > 10 g/dL Serum calcium normal On roentgenogram, normal bone structure or solitary bone plasmacytoma only Low M-component production rates (IgG value < 5 g/dL, IgA value < 3 g/dL, Bence Jones protein < 4 g/24h) Stage II: Overall data as minimally abnormal for stage I, and no single value as abnormal as defined for stage III Stage III: 1 or more of below: Hemoglobin < 8.5 g/dL Serum calcium > 12 mg/dL Advanced lytic bone lesions (scale 3) High-M-component production rates (IgG value > 7 g/dL, IgA value > 5 g/dL, Bence Jones protein > 12 g/24h)
  participants
    Stage I | 7
    Stage II | 16
    Stage III | 13
Eastern Cooperative Oncology Group Performance Status] (ECOG) [Number; unit: participants] — The ECOG scale is as follows: Grade 0: Fully active, able to carry on all pre-disease activities without restriction; Grade 1: Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature; Grade 2: Ambulatory and capable of all self-care but unable to work. Up and about more than 50% of waking hours; Grade 3: Capable of only limited self-care, confined to bed or chair > 50% of waking hours; Grade 4: Completely disabled. Cannot carry on any self-care. Confined to bed or chair.
  participants
    0 = (Asymptomatic) | 17
    1 = (Symptomatic but completely ambulatory) | 16
    2 = (Ambulatory but unable to work) | 3
    3 = (Limited self-care) | 0
    4 = (Completely disabled) | 0
Prior Chemotherapy Regimens [Median (Full Range); unit: regimens] — The number of prior chemotherapy regimens for myeloma
  regimens | 6.0 [2 to 14]
Prior Stem Cell Transplant for Myeloma [Number; unit: participants]
  Yes | 19
  No | 17
Durie-Salmon Multiple Myeloma staging at screening [Number; unit: participants] — Stages are: Stage I: Hemoglobin > 10 g/dL Serum calcium normal On roentgenogram, normal bone structure or solitary bone plasmacytoma only Low M-component production rates (IgG value < 5 g/dL, IgA value < 3 g/dL, Bence Jones protein < 4 g/24h) Stage II: Overall data as minimally abnormal for stage I, and no single value as abnormal as defined for stage III Stage III: 1 or more of below: Hemoglobin < 8.5 g/dL Serum calcium > 12 mg/dL Advanced lytic bone lesions (scale 3) High-M-component production rates (IgG value > 7 g/dL, IgA value > 5 g/dL, Bence Jones protein > 12 g/24h)
  participants
    Stage I | 7
    Stage II | 16
    Stage III | 13

OUTCOME MEASURES:

1. Primary Outcome: Myeloma Response Rate Based on the International Myeloma Working Group (IMWG) Uniform Response Criteria
Description: Myeloma response was defined as a best overall response of stringent complete response (SCR), complete response (CR), very good partial response (VGPR) or partial response (PR) SCR: CR and normal free light chain (FLC) ratio and no clonal cells in bone marrow; CR: Negative serum and urine on immunofixation, disappearance of any soft tissue plasmacytomas and ≤ 5% plasma cells in bone marrow; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥ 90% reduction in serum M-protein and urine M-protein level < 100 mg/24 hours; PR: ≥ 50% reduction of serum M-Protein and reduction in urinary M-protein by ≥ 90% or to < 200 mg/24 hours. In addition to the above, if present at baseline a ≥ 50% reduction in the size of soft tissue plasmacytomas is also required.
Time Frame: From the first dose until the data cut-off date of 03 Sept 2014; Maximum time in follow-up was 36.0 weeks.
Population: Efficacy Evaluable Population includes all participants who met eligibility criteria, took at least one dose of study medication, and had a baseline and a post-baseline efficacy assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants responding
Groups:
- Pomalidomide Plus Dexamethasone: Participants received 4 mg pomalidomide administered by mouth on Days 1-21 of each 28-day treatment cycle and 40 mg dexamethasone (participants > 75 years of age received 20 mg dexamethasone) administered by mouth once per day on Days 1, 8, 15, and 22 of a 28-day cycle until disease progression.
Arm/Group | Pomalidomide Plus Dexamethasone
Number analyzed (Participants) | 36
percentage of participants responding | 25.0 [10.855 to 39.145]
Statistical Analysis 1: Comparison: Pomalidomide Plus Dexamethasone; Test type: Superiority or Other; p = 0.0027, Binomial test for dichotomized response — Based on one sample binomial test for dichotomized response proportion against the null hypothesis(H0: p = 0.1)

2. Secondary Outcome: Myeloma Response Rate Based on European Group for Blood and Marrow Transplantation (EBMT) Criteria
Description: Myeloma response was defined as a best overall response of complete response (CR) or partial response (PR) CR is defined as: - Absence of original monoclonal paraprotein in serum and urine by immunofixation maintained at least 42 days. - <5% plasma cell in bone marrow aspirate and on bone marrow biopsy, if performed. - No increase in size or number of lytic bone lesions. - Disappearance of soft tissue plasmacytomas. PR requires all of the following: - ≥ 50% reduction in level of serum monoclonal paraprotein, maintained at least 42 days. - Reduction in 24-hour urinary light chain extraction by ≥ 90% or to < 200 mg, maintained at least 42 days. - For patients with non-secretory myeloma, ≥ 50% reduction in plasma cells in bone marrow aspirate and on biopsy, if performed, for at least 42 days. - ≥ 50% reduction in the size of soft tissue plasmacytomas. - No increase in size or number of lytic bone lesions.
Time Frame: From first dose until the data cut-off date of 03 September 2014; maximum time in follow-up was 36.0 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants responding
Arm/Group | Pomalidomide Plus Dexamethasone
Number analyzed (Participants) | 36
percentage of participants responding | 22.2 [8.642 to 35.803]

3. Secondary Outcome: Time to Response
Description: Time to response was calculated as the time from the first dose to the initial documented response (partial response or better) based on IMWG criteria. SCR: CR and normal free light chain (FLC) ratio and no clonal cells in bone marrow; CR: Negative serum and urine on immunofixation, disappearance of any soft tissue plasmacytomas and ≤ 5% plasma cells in bone marrow; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥ 90% reduction in serum M-protein and urine M-protein level < 100 mg/24 hours; PR: ≥ 50% reduction of serum M-Protein and reduction in urinary M-protein by ≥ 90% or to < 200 mg/24 hours. If present at baseline a ≥ 50% reduction in size of soft tissue plasmacytomas is also required.
Time Frame: From the first dose until the data cut-off date of 03 September 2014. Maximum time on follow-up was 36.0 weeks.
Population: Included participants with at least a PR or better based on Assessment using IMWG criteria.
Measure: Median (Full Range); unit: weeks
Arm/Group | Pomalidomide Plus Dexamethasone
Number analyzed (Participants) | 9
weeks | 4.10 [4.10 to 24.1]

4. Primary Outcome: Myeloma Response Rate Based on the International Myeloma Working Group (IMWG) Uniform Response Criteria (Later Cut-off Date)
Description: as for outcome 1
Time Frame: From the first dose until the final data cut-off date of 25 September 2015; maximum duration on treatment was 80.9 weeks
Population: Efficacy Evaluable Population (EEP) includes all participants who met eligibility criteria, took at least one dose of study medication, and had a baseline and a post-baseline efficacy assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants responding
Arm/Group | Pomalidomide Plus Dexamethasone
Number analyzed (Participants) | 36
percentage of participants responding | 41.7 [25.562 to 57.771]

5. Secondary Outcome: Myeloma Response Rate Based on European Group for Blood and Marrow Transplantation (EBMT) Criteria (Later Cut-off Date)
Description: as for outcome 2
Time Frame: as for outcome 4
Population: EEP includes all participants who met eligibility criteria, took at least one dose of study medication, and had a baseline and a post-baseline efficacy assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants responding
Arm/Group | Pomalidomide Plus Dexamethasone
Number analyzed (Participants) | 36
percentage of participants responding | 38.9 [22.964 to 54.814]

6. Secondary Outcome: Time to Response (Later Cut-off Date)
Description: as for outcome 3
Time Frame: as for outcome 4
Population: Included participants with at least a PR or better based on Assessment using IMWG criteria; EPP includes all participants who meet eligibility criteria, take at least one dose of study medication, and have a baseline and a post-baseline efficacy assessment.
Measure: Median (Full Range); unit: weeks
Arm/Group | Pomalidomide Plus Dexamethasone
Number analyzed (Participants) | 15
weeks | 8.10 [4.1 to 24.1]

7. Secondary Outcome: Kaplan-Meier Estimates of Duration of Response
Description: Duration of response (calculated for responders only) was defined as time from the initial documented response (partial response or better) to confirmed disease progression, based on IMWG criteria.
Time Frame: From first dose until the data cut-off date of 03 September 2014; maximum time for follow-up was 36 weeks
Population: Duration of Response was not analyzed as there was insufficient data available at Cycle 2, Day 1 of study treatment. There was limited data evaluated and data were not analyzed.
Arm/Group | Pomalidomide Plus Dexamethasone
Number analyzed (Participants) | 0

8. Secondary Outcome: Kaplan-Meier Estimates of Duration of Response (Later Cut-off Date)
Description: as for outcome 7
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pomalidomide Plus Dexamethasone
Number analyzed (Participants) | 15
weeks | NA [20.100 to NA] — The median duration of response based on Kaplan-Meier estimate had not been reached. The upper limit was not calculable because an insufficient number of participants reached the event at the time point for the assessment.

9. Secondary Outcome: Kaplan-Meier Estimates of Progression-free Survival (PFS)
Description: PFS was calculated as the time from the first dosing to the first documented progressive disease, as determined by the investigators based on the IMWG Uniform Response criteria, or death, whichever occurred earlier
Time Frame: From the first dose until the data cut-off date of 03 September 2014; maximum time on treatment was 36.0 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pomalidomide Plus Dexamethasone
Number analyzed (Participants) | 36
weeks | 19.0 [8.100 to NA] — The upper limit was not calculable because an insufficient number of participants reached the event at the time point for assessment

10. Secondary Outcome: Kaplan-Meier Estimates of PFS (Later Cut-off Date)
Description: as for outcome 9
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pomalidomide Plus Dexamethasone
Number analyzed (Participants) | 36
weeks | 32.10 [9.700 to NA] — The upper limit was not calculable because an insufficient number of participants reached the event at the time point for the assessment.

11. Secondary Outcome: Number of Participants With Adverse Events
Description: Relation to study drug was assessed by the Investigator as either suspected or not suspected. Counts represent the suspected relationship. Severity was assessed using National Cancer Institute Common Toxicity Terminology Criteria for Adverse Events version 4.0 (NCI CTCAE v4.0): 1= Mild 2= Moderate 3= Severe 4= Life-threatening and 5= Death related to AE. Serious AEs (SAEs) were those that resulted in death, were life-threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant disability/incapacity, congenital anomaly, or resulted in an important medical event that may have jeopardized the patient or required medical or surgical intervention to prevent one of the outcomes listed above. Treatment Emergent Adverse Event (TEAE) was defined as any AE occurring on or after the first treatment of the study medication and within 28 days after the last dose.
Time Frame: From first dose of study drug to final data cut-off date of 25 Sept 2015, maximum duration on treatment was 80.9 weeks
Population: Safety population includes all participants who took at least one dose of study medication.
Measure: Number; unit: participants
Groups:
- Pomalidomide Plus Dexamethasone: Participants received 4 mg pomalidomide administered by mouth on Days 1-21 of each 28-day treatment cycle and 40 mg dexamethasone (participants > 75 years of age received 20 mg dexamethasone) administered by mouth once per day on Days 1, 8, 15, and 22 of a 28-day cycle until disease progression or pomalidomide discontinuation for any reason.
Arm/Group | Pomalidomide Plus Dexamethasone
Number analyzed (Participants) | 36
participants
  Any 1 TEAE | 36
  TEAE related to any study drugs | 33
  TEAE related to Pomalidomide | 33
  TEAE related to Dexamethasone(Dex) | 27
  TEAE with ≥ Grade (GR) 3 | 33
  ≥ 1TEAE ≥ GR 3 related to any study drug | 30
  TEAE ≥ GR 3 related to Pomalidomide | 30
  TEAE ≥ GR 3 related to Dexamethasone | 11
  ≥ 1 serious TEAE | 16
  Serious TEAE related to any study drug | 8
  Serious TEAE related to Pomalidomide | 8
  Serious TEAE related to Dexamethasone | 6
  TEAE leading to stopping of any study drug | 5
  TEAE leading to discontinuation of Pomalidomide | 5
  TEAE leading to discontinuation of Dexamethasone | 5
  Related TEAE leading to stopping of study drug | 4
  Related TEAE leading to stopping of Pomalidomide | 4
  Related TEAE leading to stopping Dexamethasone | 4
  TEAE leading to dose reduction of any study drug | 19
  TEAE leading to dose reduction of Pomalidomide | 10
  TEAE leading to dose reduction of Dexamethasone | 15
  TEA leading to dose interruption of any study drug | 20
  TEAE leading to dose interruption of Pomalidomide | 18
  TEAE leading to dose interruption of Dexamethasone | 11
  Related TEAE leading to dose reduction of any drug | 18
  Related TEAE causing a dose reduction Pomalidomide | 10
  ≥1 related TEAE causing a dose reduction: Dex | 14
  Related TEAE leading to interruption of drugs | 16
  Related TEAE causing an interruption Pomalidomide | 15
  Related TEAE causing an interruption to Dex | 8
  TEAE Grade 5 | 3

ADVERSE EVENTS:
Time Frame: From the start of study drug through 28 days after the last dose of study drug. Maximum duration of study treatment was 80.9 weeks; up to 25 September 2015 data cut-off
Arm/Group | Pomalidomide Plus Dexamethasone
Serious Adverse Events (participants affected / at risk) | 16/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pomalidomide Plus Dexamethasone (N=36)
ANAEMIA (Blood and lymphatic system disorders) | 5
NEUTROPENIA (Blood and lymphatic system disorders) | 2
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1
PNEUMONIA (Infections and infestations) | 5
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 2
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1
MULTI-ORGAN FAILURE (General disorders) | 1
PYREXIA (General disorders) | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
CONSTIPATION (Gastrointestinal disorders) | 2
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1
BLOOD FIBRINOGEN DECREASED (Investigations) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
URINARY RETENTION (Renal and urinary disorders) | 1
SHOCK HAEMORRHAGIC (Vascular disorders) | 1
BRONCHITIS (Infections and infestations) | 1
MENINGITIS (Infections and infestations) | 1
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 1
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1
C-REACTIVE PROTEIN INCREASED (Investigations) | 1
CARDIAC FAILURE (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pomalidomide Plus Dexamethasone (N=36)
NEUTROPENIA (Blood and lymphatic system disorders) | 26
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 16
ANAEMIA (Blood and lymphatic system disorders) | 17
LYMPHOPENIA (Blood and lymphatic system disorders) | 8
LEUKOPENIA (Blood and lymphatic system disorders) | 6
PYREXIA (General disorders) | 9
OEDEMA PERIPHERAL (General disorders) | 7
MALAISE (General disorders) | 6
FATIGUE (General disorders) | 4
CONSTIPATION (Gastrointestinal disorders) | 9
DIARRHOEA (Gastrointestinal disorders) | 7
NAUSEA (Gastrointestinal disorders) | 7
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2
HAEMORRHOIDS (Gastrointestinal disorders) | 2
PROCTALGIA (Gastrointestinal disorders) | 2
VOMITING (Gastrointestinal disorders) | 2
RASH (Skin and subcutaneous tissue disorders) | 7
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 3
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 2
NASOPHARYNGITIS (Infections and infestations) | 9
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4
BRONCHITIS (Infections and infestations) | 2
PNEUMONIA (Infections and infestations) | 3
DECREASED APPETITE (Metabolism and nutrition disorders) | 4
HYPERURICAEMIA (Metabolism and nutrition disorders) | 4
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 4
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 2
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 2
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 3
DYSGEUSIA (Nervous system disorders) | 5
HYPERSOMNIA (Nervous system disorders) | 2
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2
SOMNOLENCE (Nervous system disorders) | 2
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 4
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 3
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 2
ANXIETY (Psychiatric disorders) | 3
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 3
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 3
HERPES ZOSTER (Infections and infestations) | 3
CYSTITIS (Infections and infestations) | 2
GASTROENTERITIS (Infections and infestations) | 2
DIABETES MELLITUS (Metabolism and nutrition disorders) | 2
INSOMNIA (Psychiatric disorders) | 6
RESTLESSNESS (Psychiatric disorders) | 2
INCREASED APPETITE (Metabolism and nutrition disorders) | 2
HEADACHE (Nervous system disorders) | 2
NEUROPATHY PERIPHERAL (Nervous system disorders) | 2
TREMOR (Nervous system disorders) | 2
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2
WEIGHT DECREASED (Investigations) | 2
WEIGHT INCREASED (Investigations) | 2
HYPOTENSION (Vascular disorders) | 2
HYPOTHYROIDISM (Endocrine disorders) | 2
HYPOGAMMAGLOBULINAEMIA (Immune system disorders) | 2
Pharyngitis (Infections and infestations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure agreements varied; the Investigators shall not disclose any material/information disclosed by the Sponsor (Celgene KK) with the clinical trial or information obtained by conducting the clinical trial to third parties without Sponsor's prior written approval.